CLINICAL TRIAL: NCT07026643
Title: Auricular Vagal Neuromodulation Therapy in Postural Orthostatic Tachycardia Syndrome: Physiological Mechanisms and Systemic Effects - A Pilot Study
Brief Title: aVNT in POTS - Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB25-1014
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS)
Keywords: Postural Orthostatic Tachycardia Syndrome; Auricular vagal neuromodulation therapy
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Intervention Model Description: Patients in both groups will receive daily stimulation with the Parasym device, temporarily connected to the tragus of the right ear. The stimulation parameters will be frequency of 20 Hz, pulse width of 200 µs, and the stimulation amplitude will be titrated to 1 mA below the discomfort threshold, consistent with parameters used in published clinical studies.54-56 With this stimulation at just below the discomfort threshold, people will often feel the stimulation for less than 60 seconds before they lose awareness of the ongoing stimulation. The stimulation will continue for 1 hour daily for 3 months, and we will track its use with a patient diary. Participants can continue their regular activities while wearing the aVNT device, as long as it is not soaked in water. Parasym will obtain Health Canada approval for use of their device in the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be performed on the day of the baseline evaluation before giving the participant their aVNT device. To minimize concealment bias, variable block randomization (blocks of 4 or 6) will be used. The site will access the central RedCap randomization module to determine the assignment from the randomization tables. An unblinded coordinator at the site will perform the randomization and deliver the aVNT (with appropriate programming) to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active aVNT (Experimental): For rigorous mechanistic evaluation and to establish causal relationships, intervention strategies (active aVNT vs. Sham) will be randomized among participants in this mechanistic study, ensuring that observed physiological effects are attributable to aVNT rather than placebo effects, baseline variability, or confounding factors. Patients with POTS will be randomly assigned to 3 months of active aVNT or sham treatment in 1:1 ratio. Patients will continue their stable ongoing non-pharmacological and pharmacological treatments for POTS. We will perform in-laboratory evaluations at baseline and 3 months post-randomization. We will also collect data on HR and orthostatic tachycardia at home in between the laboratory evaluations, using a wearable monitor.
  Interventions: Device: active aVNT vs. Sham
- Sham (Experimental): For rigorous mechanistic evaluation and to establish causal relationships, intervention strategies (active aVNT vs. Sham) will be randomized among participants in this mechanistic study, ensuring that observed physiological effects are attributable to aVNT rather than placebo effects, baseline variability, or confounding factors. Patients with POTS will be randomly assigned to 3 months of active aVNT or sham treatment in 1:1 ratio. Patients will continue their stable ongoing non-pharmacological and pharmacological treatments for POTS. We will perform in-laboratory evaluations at baseline and 3 months post-randomization. We will also collect data on HR and orthostatic tachycardia at home in between the laboratory evaluations, using a wearable monitor.
  Interventions: Device: active aVNT vs. Sham

INTERVENTIONS:
Device: active aVNT vs. Sham — Patients in both groups will receive daily stimulation with the Parasym device, temporarily connected to the tragus of the right ear (Fig 2).54 The stimulation parameters will be frequency of 20 Hz, pulse width of 200 µs, and the stimulation amplitude will be titrated to 1 mA below the discomfort threshold, consistent with parameters used in published clinical studies.54-56 With this stimulation at just below the discomfort threshold, people will often feel the stimulation for less than 60 seconds before they lose awareness of the ongoing stimulation. The stimulation will continue for 1 hour daily for 3 months, and we will track its use with a patient diary. Participants can continue their regular activities while wearing the aVNT device, as long as it is not soaked in water. Parasym will obtain Health Canada approval for use of their device in the study.

SUMMARY:
Autonomic nervous system imbalance causes postural tachycardia and related cardiac symptoms in Postural Orthostatic Tachycardia Syndrome (POTS). The impact of POTS is more far-reaching than postural tachycardia. Several systemic, autonomic symptoms along with neuro-cognitive dysfunction leading to poor quality of life contribute to significant disability in POTS. A combination of abnormal autonomic tone, abnormal cerebral blood flow regulation, and systemic inflammation may contribute to POTS symptoms.

Auricular Vagal Neuromodulation Therapy (aVNT) has the potential for multisystem holistic benefit for patients with POTS: Autonomic neuromodulation by aVNT might address multiple aspects of POTS pathophysiology and improve POTS symptoms. It can reduce postural tachycardia by increasing the parasympathetic (PNS) and decreasing sympathetic (SNS) tone. In patients undergoing vagus nerve stimulation for various indications, an increase in PNS tone has been associated with improved middle cerebral artery velocity (MCAv) at rest and during cognitive stress. aVNT has been associated with improved cerebral blood flow and reduced infarct size in an experimental model of ischemic stroke, suggesting similar improvements in cerebral autoregulation in POTS. Vagus nerve stimulation has also been linked to improved cognitive function. The anti-inflammatory effect and improved endothelial function might improve cerebral blood flow regulation and cognitive function. The anti-inflammatory effects of aVNT may improve postural hemodynamics, reduce postural tachycardia, relieve other POTS symptoms, and improve quality of life (QoL). POTS is a complex multisystem disorder with debilitating symptoms that currently lack effective treatments. aVNT has the potential to recalibrate autonomic tone dysregulation, enhance MCAv, improve cognitive function, reduce inflammation, and ultimately improve symptoms and quality of life in POTS patients.

DETAILED DESCRIPTION:
Postural Orthostatic Tachycardia Syndrome (POTS) is a chronic disorder characterized by dysregulation of the cardiovascular autonomic nervous system, leading to an excessive increase in heart rate upon standing. The pathophysiology of POTS is multifactorial, involving systemic inflammation, dysfunctional autonomic modulation, cerebral hypoperfusion, and impaired cerebral autoregulation. Beyond the hallmark postural tachycardia, POTS is associated with numerous systemic, autonomic, and neurocognitive symptoms that severely impair quality of life (QoL). Current treatments for POTS are limited in number, tolerability, efficacy, and evidence base.1, 2 Auricular vagal neuromodulation therapy (aVNT), a noninvasive method of vagus nerve stimulation, has shown potential due to its autonomic neuromodulation and anti-inflammatory effects. The global hypothesis is that autonomic dysregulation and systemic inflammation underlie POTS and its chronic symptoms. We will test this hypothesis using the neuromodulation effects of chronic, intermittent aVNT in patients with POTS to restore autonomic balance and reduce systemic inflammation leading to improved hemodynamics cognition and symptoms. We will test this hypothesis with a sham-controlled, double-blind, randomized mechanistic study of aVNT in 80 patients with POTS.

POTS is a chronic, multisystem disorder with symptomatic orthostatic intolerance and an excessive increase in heart rate (HR) upon standing without significant orthostatic hypotension (Fig 1). Patients often have low cardiac filling pressures and low stroke volume that worsens with upright posture. These lead to symptoms such as palpitations, low energy, headaches, cognitive impairment, muscle fatigue, chest pain, and generalized weakness. POTS is a debilitating autonomic nervous system disorder affecting ~1% of the population (~400,000 Canadians).

POTS predominantly affects females, with a female-to-male ratio of 5:1. The impact of POTS is particularly significant because it affects adolescent and young adult females who are typically in critical stages of their education or early careers. This often leads to frequent absences from school or work and necessitates lifestyle adjustments that hinder social and professional opportunities. POTS delays/limits their education, and leads to both direct and indirect economic loss. Consequently, POTS presents a considerable public health challenge with extensive social and economic implications, given its effect on a predominantly young and productive segment of the population.

Our research considers POTS holistically, with research priorities developed through a partnered research approach. Our patient partners, including Dysautonomia International, have long prioritized consideration of symptoms and outcomes beyond orthostatic tachycardia. POTS patients frequently experience several noncardiac symptoms including low energy, fatigability, and anxiety. Most POTS patients suffer from sleep disturbances, and mild to moderate depression is common. Symptoms related to subjective cognitive dysfunction, often referred to as "brain fog", are disabling and reported by over >90% of patients with POTS. Many systemic, autonomic, and neurocognitive symptoms occur even when supine, but are worse with upright posture. Severe fatigue, sleep disturbances, and "brain fog" are reported in >90% of patients with POTS. These noncardiac symptoms of POTS are often debilitating, severely affecting daily functioning, and reducing quality of life (QoL) to levels comparable to patients with heart failure.

Many POTS patients report cognitive dysfunction and mental fatigue, experiencing symptoms that significantly impair intellectual functioning and interfere with daily activities. A questionnaire-based study revealed that over 95% of POTS patients reported cognitive impairment, with many experiencing daily symptoms, including difficulties with executive function. These cognitive deficits are comparable to those observed in chronic fatigue syndrome and multiple sclerosis, indicating their severity and impact. Cognitive dysfunction can occur even while lying down or seated. In our prior study of 28 female POTS patients and 24 matched healthy controls, significant reductions in selective attention, cognitive processing speed, and executive function were observed, indicating that tasks requiring planning, organizing, and adapting are particularly affected in POTS. Many patients report worsened symptoms when upright. Using the Cambridge Neuropsychological Test Automated Battery (CANTAB), we found that POTS patients had worse cognitive processing than controls while seated (375±9 vs. 337±18 ms, p=0.045), and more so when standing (382±18 vs. 320±11 ms, p=0.012). While the pathophysiology of cognitive impairment in POTS is not understood, decreased PNS tone has been linked to both aging-associated cognitive decline and transient cognitive impairment following orthostatic stress.

Intact cerebral autoregulation maintains constant cerebral blood flow during postural changes. In contrast, impaired cerebral autoregulation has been linked with symptoms of cognitive dysfunction in POTS. Unlike peripheral vascular beds, the cerebral vasculature is densely innervated by parasympathetic (PNS) fibers, and PNS-mediated vasodilation maintains adequate cerebral blood flow. Reduced cerebrovascular PNS activity has been linked to impaired blood flow. MCAv can be measured with transcranial Doppler. POTS patients show a significantly greater reduction in middle cerebral artery velocity (MCAv) during tilt testing compared to healthy controls. This occurs without significant hypotension, indicating impaired cerebral autoregulatory control, which could result from autonomic dysregulation. Reduced MCAv occurs in seated POTS patients during cognitive stress. POTS patients also exhibit reduced functional hyperemia and abnormal MCAv responses upon standing.

Intact cerebral autoregulation maintains constant cerebral blood flow during postural changes. In contrast, impaired cerebral autoregulation has been linked with symptoms of cognitive dysfunction in POTS. Unlike peripheral vascular beds, the cerebral vasculature is densely innervated by parasympathetic (PNS) fibers, and PNS-mediated vasodilation maintains adequate cerebral blood flow. Reduced cerebrovascular PNS activity has been linked to impaired blood flow. MCAv can be measured with transcranial Doppler. POTS patients show a significantly greater reduction in middle cerebral artery velocity (MCAv) during tilt testing compared to healthy controls. This occurs without significant hypotension, indicating impaired cerebral autoregulatory control, which could result from autonomic dysregulation. Reduced MCAv occurs in seated POTS patients during cognitive stress. POTS patients also exhibit reduced functional hyperemia and abnormal MCAv responses upon standing.

Acute viral infections (like the flu) often trigger POTS-like symptoms, including postural tachycardia, fatigue, and brain fog. While typically transient, these symptoms can lead to long-term POTS in some patients, suggesting that infection-related inflammation may be involved in its pathogenesis. Recent studies indicate that POTS is marked by low-grade inflammation, with elevated levels of pro-inflammatory cytokines such as IL-6, IL-18, IL-21, and TNFα, absent in healthy controls.

A continuous communication between ANS and the immune system maintains physiological homeostasis. The vagus nerve modulates inflammation through the inflammatory reflex. The afferent component of this reflex is activated by inflammatory cytokines, while the efferent signals from the brainstem vagal center are carried by the splenic nerve. This reflex reduces cytokine release by splenic macrophages by activating the α7 nicotinic cholinergic receptors (α7nAChR). Hence, autonomic imbalance with reduced PNS activity in POTS may contribute to this systemic pro-inflammatory state.

A continuous communication between ANS and the immune system maintains physiological homeostasis. The vagus nerve modulates inflammation through the inflammatory reflex. The afferent component of this reflex is activated by inflammatory cytokines, while the efferent signals from the brainstem vagal center are carried by the splenic nerve. This reflex reduces cytokine release by splenic macrophages by activating the α7 nicotinic cholinergic receptors (α7nAChR). Hence, autonomic imbalance with reduced PNS activity in POTS may contribute to this systemic pro-inflammatory state.

Treatments for POTS aim to expand blood volume (increased salt and water intake, fludrocortisone), minimize gravitational pooling (compression garments, midodrine), and reduce sinus rate with sympatholytic (β-blockers), parasympathomimetic (pyridostigmine), or funny channel inhibitors. While these therapies reduce postural tachycardia, there is little data on their impact on the broader spectrum of symptoms associated with POTS. They are generally ineffective for non-cardiac symptoms. Additionally, the side effects of these medications often limit their tolerability; for instance, β-blockers, especially in higher doses, pyridostigmine, and central sympatholytic agents may exacerbate noncardiac symptoms such as fatigue, gastrointestinal disturbances, drowsiness, and cognitive impairments. Although the nonspecific stimulant modafinil can improve cognitive dysfunction, it may also increase postural tachycardia. Overall, many POTS patients continue to experience significant impairment in quality of life, leaving them feeling that their condition remains inadequately managed.

aVNT is a novel, noninvasive strategy for stimulating the auricular branch of the vagus nerve at the tragus of the external ear (Fig 2; Parasym Health; https://www.parasym.co/parasym-device.html). This method selectively activates afferent fibers that project to the nucleus tractus solitarius (NTS), the primary sensory nucleus of the vagus in the brainstem. Activation of the NTS subsequently stimulates the nucleus ambiguus (NA) and the caudal ventrolateral medulla (CVLM). The activation of the NA leads to the engagement of vagal efferent fibers, while activation of the CVLM inhibits sympathetic pacemaker neurons in the rostral ventrolateral medulla. This process ultimately increases PNS tone and decreases SNS tone.

By enhancing the parasympathetic inflammatory reflex, aVNT is shown to exert systemic anti-inflammatory effects. Its anti-inflammatory properties have been demonstrated in both acute endotoxemia and chronic systemic inflammatory diseases. Additionally, aVNT has been shown to decrease inflammatory cytokines in cardiovascular diseases, including arrhythmias and heart failure. The mechanistic basis of these effects is supported by pharmacological evidence, where the administration of methyllycaconitine, an α7nAChR antagonist, attenuates the anti-inflammatory action of aVNT. This finding suggests that aVNT mediates its effects through activation of the cholinergic anti-inflammatory pathway, further reinforcing its potential therapeutic role in conditions characterized by autonomic dysregulation and systemic inflammation.

Parasym neuromodulation has been studied in different clinical disorders. Daily Parasym aVNT for 1h resulted in an 85% reduction in paroxysmal atrial fibrillation burden (p=0.01). In patients with heart failure with preserved ejection fraction, daily Parasym aVNT for 1h for three months led to significant improvements in cardiac function. In a pilot study in acute decompensated heart failure, twice daily aVNT led to a significant reduction in systemic inflammation (IL-6 ↓78% vs. 9%; p=0.012), and attenuation of oxidative stress.

Parasym aVNT has consistently demonstrated autonomic neuromodulatory effects and systemic anti-inflammatory effects (↓TNF-α, ↓IL-6) across studies. Prior trials of Parasym aVNT have shown that low-level tragus electrical stimulation does not acutely induce vagotonia or sinus bradycardia. Over a few months, this therapy is safe and well-tolerated, with no significant adverse effects.

Invasive vagus nerve stimulation has been widely used for refractory epilepsy, with anecdotal reports suggesting improvement in orthostatic symptoms in patients with concurrent POTS. Early investigations into vagal neuromodulation for POTS demonstrated that short-term aVNT during tilt testing reduced postural tachycardia, providing initial evidence of its autonomic effects. An open-label study involving daily aVNT for 14 days demonstrated a significant reduction in orthostatic intolerance and gastrointestinal symptoms in POTS patients, with a trend towards a reduced heart rate upon standing also observed in the aVNT group. A recent randomized, sham-controlled trial by Stavrakis et al evaluated chronic aVNT in POTS using the Parasym device. The study enrolled 26 patients who received one hour of daily aVNT (n=12) or sham stimulation (n=14) for two months. aVNT significantly reduced postural tachycardia (17.6±9.9 bpm vs. 31.7±14.4 bpm; p=0.01) without inducing orthostatic hypotension, suggesting improved heart rate regulation. Wang et al. found that aVNT daily for one-hour sessions over one month significantly attenuated postural tachycardia in patients with POTS following COVID-19 infection, with enhanced cardiovagal function during heart rate variability analysis. None of the studies, however, evaluated the impact of aVNT on POTS symptoms, cognitive function, or cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* POTS Patients: POTS patients will meet Canadian Cardiovascular Society criteria. 6 POTS patients will have orthostatic tachycardia >30 bpm increase in HR within 10 minutes of upright posture [>40 bpm in patients <20 years]), in the absence of orthostatic hypotension (drop in BP >20/10 mmHg), chronic symptoms of orthostatic intolerance, and no obvious cause for the tachycardia.
* Age between 18-80 years
* Male and female subjects are eligible
* Able and willing to provide informed consent

Exclusion Criteria:

* Unable to give informed consent
* Stimulant use within one week of the study
* Systolic blood pressure >150 mm Hg and/or diastolic blood pressure > 100 mm Hg
* Neurogenic orthostatic hypotension, prior stroke, myocardial infarction or heart failure, hematocrit < 28%
* Significant comorbidities (cardiovascular, metabolic, renal, respiratory, cancer, immunological or hematological)
* History of vagotomy, permanent pacemakers
* Pregnant or nursing females.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic aVNT in POTS induces favorable autonomic neuromodulation and decreases orthostatic tachycardia | We will perform in-laboratory evaluations at baseline and 3 months post-randomization.
  For rigorous mechanistic evaluation and to establish causal relationships, intervention strategies (active aVNT vs. Sham) will be randomized among participants in this mechanistic study, ensuring that observed physiological effects are attributable to aVNT rather than placebo effects, baseline variability, or confounding factors. Patients with POTS will be randomly assigned to 3 months of active aVNT or sham treatment in 1:1 ratio.
chronic aVNT in POTS induces favorable autonomic neuromodulation and decreases orthostatic tachycardia | We will perform in-laboratory evaluations at baseline and 3 months post-randomization.
  For rigorous mechanistic evaluation and to establish causal relationships, intervention strategies (active aVNT vs. Sham) will be randomized among participants in this mechanistic study, ensuring that observed physiological effects are attributable to aVNT rather than placebo effects, baseline variability, or confounding factors. Patients with POTS will be randomly assigned to 3 months of active aVNT or sham treatment in 1:1 ratio. Patients will continue their stable ongoing non-pharmacological and pharmacological treatments for POTS.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Raj, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: Undecided